CLINICAL TRIAL: NCT07234851
Title: SYNAPSING's POSTMORTEM AND IN VITRO STUDIES OF SYNAPSE DYSFUNCTION
Brief Title: Understanding Mechanisms of Synaptic Degeneration Underlying Clinical Symptoms in Patients With MDs and NDs.
Status: Enrolling by invitation | Type: Observational
Sponsor: Fundació Institut de Recerca de l'Hospital de la Santa Creu i Sant Pau (Other)
Collaborators: University of Eastern Finland (Other); University of the Basque Country (UPV/EHU) (Other); Natural and Medical Sciences Institute (NMI) (Unknown)
Responsible Party: Sponsor
Other Study IDs: IIBSP-NCP-2024-174
Record Dates: First submitted 2025-03-17; First posted 2025-11-19 (Actual); Last update posted 2025-12-11 (Actual); Status verified 2025-11

CONDITIONS: Schizophrenia Disorder; Frontotemporal Dementia, Behavioral Variant; Major Depressive Disorder (MDD); Bipolar Disorder (BD); Alzheimer's Disease
Keywords: synapse; biomarker; induced pluripotent stem cells; mental disorder; neurodegenerative disorder; biofluids; psychiatric symptoms
MeSH Terms: conditions — Schizophrenia; Pick Disease of the Brain; Depressive Disorder, Major; Bipolar Disorder; Alzheimer Disease; Mental Disorders; Neurodegenerative Diseases

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — brain tissue from necropsy, iPSC clones
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (6):
- Major depressive disorder: Cases that arrive to autopsy with a previous clinical diagnosis of major depressive disorder
- Schizophrenia: Cases that arrive to autopsy with a previous clinical diagnosis of schizophrenia or iPSC clones derived from a patient with a previous clinical diagnosis of schizophrenia
- Bipolar disorder: Cases that arrive to autopsy with a previous clinical diagnosis of major depressive disorder
- Control: Cases that arrived to autopsy without a prior diagnosis of a neurodegenerative or psychiatric condition or iPSC clones derived from a cognitively unimpaired healthy volunteer
- Alzheimer's disease: Cases that arrive to autopsy with neuropathological confirmation of Alzheimer's disease
- frontotemporal dementia: Cases that arrive to autopsy with neuropathological confirmation of frontotemporal lobar degeneration

SUMMARY:
Clinical Study A. Retrospective Neuropathological Study of Synapse dysfunction.

This is a cross-sectional study of patients retrospectively collected from existing postmortem collections and from existing collections of iPSC-derived neurons. Postmortem tissue and iPSC-derived neurons from age and sex-matched unaffected volunteers without a MD or ND diagnosis are used as controls.

DETAILED DESCRIPTION:
This study will:

1. perform RNA sequencing of postmortem synapses from the prefrontal cortex of patients with schizophrenia or frontotemporal dementia and unaffected controls. The data will be combined with already available RNA sequencing data from established iPSC clones from schizophrenia or behavioural variant frontotemporal dementia patients and unaffected controls. The postmortem frontotemporal dementia samples have already been characterised in terms of frontal cortex pathology in a previous study and data from RNA sequencing of homogenates is available for comparison. The prefrontal cortex has been implicated as a core affected region across MDs and NDs making this the perfect region to determine common molecular drivers of synapse dysfunction. Pathway analysis of the RNA sequencing dataset will be performed to identify biological pathways or individual genes that are deregulated in the postmortem samples and iPSC lines from each condition. A total of 3 genes that converge between the postmortem and iPSC datasets will be selected for gene-editing. Each gene will be CRISPR/Cas9-repaired in 1 selected schizophrenia parental line and 1 selected frontotemporal dementia parental line. The impact of the induced transcriptional changes on functional and synaptic morphology phenotypes in neuronal cultures from each gene-edited line will be compared to the respective parental line and to lines from 3 healthy controls. A rescue of the disease phenotypes is expected such that the repaired edited line shows activity and synaptic morphology comparable to the healthy control lines and distinct from the unedited parental line. All experiments will include 3 biological replicates taking the total number of analyses to 420. The study will also determine the role of microglia on neuronal deficits in iPSC-derived neurons from the 20 available clones from patients with schizophrenia or behavioural variant frontotemporal dementia by comparing electrophysiological activity and synapse morphology in iPSC-derived neurons culture alone to those observed in iPSC-derived neurons co-cultured with iPSC-derived microglia differentiated from the same clones.
2. compare the molecular composition of postmortem synapses from the prefrontal cortex across 3 MDs (major depressive disorder, bipolar disorder and schizophrenia) and identify differentially expressed proteins and dysfunctional protein networks through pathway analyses. To determine the potential effects of psychotropic drugs on synaptic proteomes, the study will quantify the concentrations of >200 psychoactive drugs and metabolites in both blood and cerebellum postmortem samples from the same donors and determine the correlation with the differentially expressed proteins. While blood analyses provide information on drugs present at the time of death, toxicological data in brain tissue, which accumulates drugs for weeks or even months after the last intake, serves as a better indicator of subjects' adherence to the treatments. Groups larger than 15 subjects are recommended for proteomic studies such as this. Each subject was paired to a control subject, matching sex, age, and postmortem interval and with no evidence of psychiatric or neurological conditions, according to their medical records.
3. quantify and compare synapse loss in brain regions shown to be associated with reduced volumes in MD and ND patients postmortem. Specifically, the study will compare synapse density in the prefrontal cortex, hippocampus and striatum from patients with major depressive disorder, bipolar disorder, schizophrenia, Alzheimer's disease, frontotemporal dementia to age and sex-matched unaffected controls.

ELIGIBILITY:
Inclusion criteria for psychiatric disorders:

* Age group: Midlife brain donors (age-at-death>40).
* Sex distribution: % Female in schizophrenia (23%), major depressive disorder and controls (40%), bipolar disorder and controls (55%). These percentages match those typically found in these disorders.
* Antemortem diagnosis of schizophrenia (paranoid-subtype diagnoses only to minimise the impact of potential confounding factors on the results and ensure homogeneity across schizophrenia subjects), major depression or bipolar disorder. Diagnoses are confirrmed antemortem by a psychiatrist using Diagnostic and Statistical Manual of Mental Disorders, fourth edition (DSM-IV) criteria, as recorded in the deceased individuals' medical records.

Exclusion criteria for psychiatric disorders:

For schizophrenia, cases displaying additional neurological or psychiatric conditions, such as histories of substance use disorder will be excluded. Postmortem delay >24h (to minimise perimortem confounding variables potentially affecting tissue quality.

Inclusion criteria for Neurodegenerative diseases:

* Age group: Latelife brain donors (age-at-death>50).
* Sex distribution: Alzheimer's disease (60%), frontotemporal dementia (65%). These percentages match those typically found in these diseases.
* Neuropathological confirmation of Alzheimer's disease or frontotemporal lobar degeneration (C9orf72 repeat expansion carrier)Alzheimer's disease

Exclusion criteria for Neurodegenerative diseases:

Postmortem delay >24h (to minimise perimortem confounding variables potentially affecting tissue quality.

Min Age: 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Resource 1. Frozen samples and paraffin sections from necropsy tissue will be provided by the University of Basque Country, Bilbao. Autopsies are performed in the Basque Institute of Legal Medicine, Bilbao, Spain.
  Resource 2. Frozen samples and paraffin sections from necropsy tissue are recruited from the neurological tissue bank collection (IDIBAPS, Barcelona).
  Resource 3. A collection of human induced pluripotent stem cell clones from clinically and genetically well-phenotyped schizophrenia (Natural and Medical Sciences Institute), behavioural variant frontotemporal dementia patients (University of Eastern Finland) and unaffected controls (both sites) that have already been functionally characterised in previous studies.
Sampling Method: Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2025-02-01 (Actual); Primary Completion 2029-06-30 (Estimated); Study Completion 2029-09-30 (Estimated)

PRIMARY OUTCOMES:
Synaptic gene dysregulation in schizophrenia and frontotemporal dementia | January 2025 to December 2029
  A list of genes that are differentially expressed in schizophrenia and frontotemporal dementia compared to controls identified by RNA sequencing a) synaptic fractions isolated from postmortem tissue from the prefrontal cortex of autopsy cases with a clinical diagnosis of schizophrenia or confirmation of frontotemporal lobar degeneration and b) established iPSC clones from patients with a clinical diagnosis of schizophrenia or behavioural variant frontotemporal dementia.
Molecular pathways related to synapse dysfunction in major depressive disorder, bipolar disorder and schizophrenia | January 2025 to December 2029
  A list of biological processes that are enriched for proteins that are differentially expressed in major depressive disorder, bipolar disorder and schizophrenia compared to controls identified by proteomic analysis of synaptic fractions isolated from postmortem tissue from the prefrontal cortex of autopsy cases with a clinical diagnosis ofmajor depressive disorder, bipolar disorder or schizophrenia
Impact of psychiatric and neurodegenerative disorders on synapse density in affected brain regions. | January 2028 to December 2029
  Density of immunoreactive objects labelled with an antibody to pre and post synapse markers (vGlut1, PSD-95) in the prefrontal cortex, hippocampus and striatum from autopsy cases with a prior diagnosis of major depressive disorder, bipolar disorder, schizophrenia and unaffected controls and brain donors with neuropathological confirmation of Alzheimer's disease or frontotemporal dementia and unaffected controls.

SECONDARY OUTCOMES:
Effects of psychotropic drugs on molecular pathways at the synapse related to major depressive disorder, schizophrenia and bipolar disorder | July 2025 to December 2027
  A list of proteins that correlate with the concentrations of >200 psychoactive drugs and metabolites in both blood and cerebellum from autopsy cases with a prior diagnosis of major depressive disorder, schizophrenia or bipolar disorder

CONTACTS AND LOCATIONS:
Locations (1):
- Research Institute Sant Pau, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: Yes
Pseudoanonymised age, biological sex, ethnicity, country of origin/residence, diagnosis, age-at-death, postmortem interval, suicide attempts, comorbidities, therapies, toxicology, synapse density, transcriptome, proteome will uploaded to Zenodo (or ProteomeXchange Consortium PRIDE repository for genomic and proteomic data), which use DOIs as persistent and unique identifiers
Supporting Information: Study Protocol, SAP, CSR, Analytic Code
Time Frame: Jan2025-Jan2035
Access Criteria: clinical and research communities